CLINICAL TRIAL: NCT04717921
Title: Can Selective Serotonin Reuptake Inhibitor Drugs Alter Retinal Nerve Fiber Layer Thickness in First Episode Depressive Patients?
Brief Title: Assesment of Retinal Nerve Fiber Layer in First Episode Depressive Patients Using Selective Serotonin Reuptake Inhibitor
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Mehmet Diyaddin Güleken (Other)
Responsible Party: Sponsor-Investigator, Mehmet Diyaddin Güleken, Medical Doctor, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Organization: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Other Study IDs: Mehmet Diyaddin Güleken
Record Dates: First submitted 2021-01-17; First posted 2021-01-22 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Unipolar Depression
Keywords: unipolar depression; optical coherence tomography; retinal nerve fiber layer; selective serotonin reuptake inhibitor
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Subjects with unipolar depression
- Healthy: Healthy Control Group

SUMMARY:
The aim of this study is to assess the changes in retinal nerve fiber layer due to SSRI treatment in first-attack major depressive patients.

DETAILED DESCRIPTION:
Selective serotonin reuptake inhibitors (SSRIs) are among the most used and safe antidepressant drugs in the world. In previous studies, SSRIs have been found to cause an increase in brain gray matter volume in patients with major depression (MD). Optical coherence tomography (OCT) is a non-invasive medical imaging method that displays biological tissue layers by taking high-resolution tomographic sections. Changes in the thickness of the retinal nerve fiber layer (RNFL), a layer of the ganglion cell complex in the retinal layer of the eye and composed of ganglion cell axons, occur due to axonal damage in the retinal nerve tissue. Since RNFL is similar to brain gray matter tissue, recently neurological and psychiatric studies have been conducted to provide data on the neurodegeneration that occurs in the brain by OCT. However, in a recent cross-sectional study, contrary to what was expected, thinning of the retinal nerve fiber layer was detected in psychiatric patients using SSRI drugs compared to the healthy group, and this was attributed to a probable maculopathy caused by SSRIs in the eye. In this study, it is aimed to assess the probable cortical volume changes of the patients by measuring the changes in retinal nerve layers due to SSRI treatment in first-attack MD patients.

ELIGIBILITY:
Inclusion Criteria:

* First attack depressive patients between 18 and 65 years
* Diagnosed with the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders 5 / Clinical Version (SCID-5 / CV)
* Started to be treated with selective serotonin reuptake inhibitors
* Having a Standardized Mini Mental Test (SMMT) score of 24 or more and
* Healthy subjects with no psychiatric history, having a SCL-90-R (GSI) score of less than 1.0

Exclusion Criteria:

* Depressive subjects with any neurological (cerebrovascular disease, head trauma, intracranial mass, dementia, epilepsy, multiple sclerosis, etc.) or general medical (such as diabetes, hypertension, myocardial infarction, etc.) diagnosis, with an ocular surgery or a history of ocular trauma, retinal pathology (detachment, etc.), other eye pathologies such as optic nerve neuropathy and refractive error, previous history of antidepressant drug use, alcohol-substance abuse or addiction,
* Healthy individuals with a history of psychiatric diagnosis or a SCL-90-R (GSI) score of 1.0 or above

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: First-episode major depressive outpatients or inpatients followed up in Psychiatry Department of Sağlık Bilimleri Üniversitesi Gazi Yaşargil Training and Research Hospital, and healthy volunteers matched with them in terms of age and gender for comparison will be included in the study.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Retinal nerve fiber layer thickness | Baseline, at first week and at the 8th week of the treatment
  Retinal nerve fiber layer thickness change during selective serotonin reuptake inhibitor treatment in first attack depressive subjects

SECONDARY OUTCOMES:
Choroid thickness | Baseline, at first week and at the 8th week of the treatment
  Choroid thickness change during selective serotonin reuptake inhibitor treatment in first attack depressive subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Sağlık Bilimleri Üniversitesi Gazi Yaşargil Tranining and Research Hospital, Diyarbakır, Turkey (Türkiye)